CLINICAL TRIAL: NCT04567810
Title: A Phase 1 Study in Healthy Participants to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single -Ascending and Multiple Doses of an Anti-Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Chicken Egg Antibody (IgY)
Brief Title: Safety, Tolerability, and Pharmacokinetics of Anti-Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Chicken Egg Antibody (IgY) (COVID-19)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: CVR001
Record Dates: First submitted 2020-09-18; First posted 2020-09-29 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Part A: 2 mg preparation (Experimental): Participants receive a single 2 mg dose of anti-SARS-CoV-2 IgY.
  Interventions: Drug: anti-SARS-CoV-2 IgY
- Part A: 4 mg preparation (Experimental): Participants receive a single 4 mg dose of anti-SARS-CoV-2 IgY.
  Interventions: Drug: anti-SARS-CoV-2 IgY
- Part A: 8 mg preparation (Experimental): Participants receive a single 8 mg dose of anti-SARS-CoV-2 IgY.
  Interventions: Drug: anti-SARS-CoV-2 IgY
- Part A: placebo preparation (Placebo Comparator): Participants receive placebo matching anti-SARS-CoV-2 IgY.
  Interventions: Drug: Placebo
- Part B: 6 mg total daily dose (Experimental): Participants receive a 2 mg dose of anti-SARS-CoV-2 IgY three times daily for 14 days.
  Interventions: Drug: anti-SARS-CoV-2 IgY
- Part B: 12 mg total daily dose (Experimental): Participants receive a 4 mg dose of anti-SARS-CoV-2 IgY three times daily for 14 days.
  Interventions: Drug: anti-SARS-CoV-2 IgY
- Part B: 24 mg total daily dose (Experimental): Participants receive a 8 mg dose of anti-SARS-CoV-2 IgY three times daily for 14 days.
  Interventions: Drug: anti-SARS-CoV-2 IgY
- Part B: 0 mg total daily dose (Placebo Comparator): Participants receive placebo matching anti-SARS-CoV-2 IgY three times daily for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: anti-SARS-CoV-2 IgY — anti-SARS-CoV-2 IgY preparation in liquid administered with a bottle with a dropper.
  Arms: Part A: 2 mg preparation; Part A: 4 mg preparation; Part A: 8 mg preparation; Part B: 12 mg total daily dose; Part B: 24 mg total daily dose; Part B: 6 mg total daily dose
Drug: Placebo — Placebo matching anti-SARS-CoV-2 IgY preparation in liquid administered with a bottle with a dropper.
  Arms: Part A: placebo preparation; Part B: 0 mg total daily dose

SUMMARY:
The primary objective of Part 1 (Single Ascending Dose) is to assess the safety and tolerability of anti-SARS-CoV-2 IgY when given as single-ascending doses administered intranasally to healthy participants.

The primary objective of Part 2 (Multiple Dose) is to assess the safety and tolerability of anti-SARS-CoV-2 IgY when given as multiple doses administered intranasally to healthy participants. A secondary objective is to assess the pharmacokinetics of anti-SARS-CoV-2 IgY when given as multiple doses administered intranasally to healthy participants.

Safety will be evaluated using adverse event (AE), physical examination (including vital signs), electrocardiogram, and clinical laboratory data. Pharmacokinetics will be evaluated by serum anti-SARS-CoV-2 IgY concentration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating females
* Body weight of at least 50 kg
* Good state of health (mentally and physically)
* Must agree to use of highly effective method of contraception

Exclusion Criteria:

* Received other investigational drug within the last 30 days prior to screening
* History of drug or alcohol abuse in the past 2 years (>21 units of alcohol per week for males and >14 units of alcohol per week for females)
* Current smoker / e-smoker
* Abnormal kidney function
* Abnormal liver function
* Positive for hepatitis B or C infection
* Positive for HIV infection
* Positive for SARS-CoV-2 infection
* History of egg allergy
* Abnormal cardiac function

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | up to 21 days

SECONDARY OUTCOMES:
Number of Participants With Vital Sign Findings Reported as TEAEs | up to 21 days
Number of Participants With Clinically Significant Findings in Physical Examinations | up to 21 days
  Clinically significant in the judgement of the investigator.
Number of Participants With Clinically Significant Changes From Baseline in ECG Data | up to 21 days
  Clinically significant in the judgement of the investigator.
Number of participants with Clinically Significant Changes from Baseline in Clinical Laboratory Parameters | up to 21 days
  Clinically significant in the judgement of the investigator.
Number of Participants with Presence of Serum anti-SARS-CoV-2 IgY | up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Daria Mochly-Rosen, PhD, Study Director — Stanford University; Michaela Lucas, MD, Principal Investigator — Linear Clinical Research
Locations (1):
- Linear Clinical Research - Harry Perkins Research Institute, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Frumkin LR, Lucas M, Scribner CL, Ortega-Heinly N, Rogers J, Yin G, Hallam TJ, Yam A, Bedard K, Begley R, Cohen CA, Badger CV, Abbasi SA, Dye JM, McMillan B, Wallach M, Bricker TL, Joshi A, Boon ACM, Pokhrel S, Kraemer BR, Lee L, Kargotich S, Agochiya M, John TS, Mochly-Rosen D. Egg-Derived Anti-SARS-CoV-2 Immunoglobulin Y (IgY) With Broad Variant Activity as Intranasal Prophylaxis Against COVID-19. Front Immunol. 2022 Jun 1;13:899617. doi: 10.3389/fimmu.2022.899617. eCollection 2022. PMID 35720389
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343